CLINICAL TRIAL: NCT07266909
Title: Impact of Attentional Tunneling or the "Tunnel Effect" in Dentistry. Multi-centre Cross-sectional Study of a Population of French Practitioners.
Brief Title: Impact of Attentional Tunelling on a Population of French Practitioners
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Odonto06
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Awareness; Attention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Public Practitioners: Practitioners working in dental departments at hospitals and university centres in Nice, Marseille and Montpellier (France)
  Interventions: Other: Face-to-face or online survey
- Orthodondics Students: Resident enrolled in France in an Orthodontics and Dentofacial Orthopedics training program, attending the national course given by the University of Nice
  Interventions: Other: Face-to-face or online survey
- Private practitioners: Private practitioners or employees (excluding university hospitals) enrolled in continuing education programmes at the university dental services in Nice, Marseille, and Montpellier (France)
  Interventions: Other: Face-to-face or online survey

INTERVENTIONS:
Other: Face-to-face or online survey — A face -to-face or online questionnaire will be given to study paticipants after a seminar on attentional tunneling organized by Professors Dridi and Charavet.

SUMMARY:
The tunnel effect, also known as attentional tunnelling, is a cognitive bias affecting all healthcare professionals, including odontologists. It is characterised by an excessive focus on a specific element of a clinical situation, which can alter the overall assessment and lead to errors in medical practice. This poses a particular risk to the quality of dental care, especially surgical care. Despite the importance of this risk, few studies have addressed this issue in dentistry. Therefore, raising the dental community's awareness of this phenomenon on a large scale is both justified and necessary.

ELIGIBILITY:
Inclusion Criteria:

* University hospital practitioner (professor, associate professor, ...)
* Dental surgeon (outside university hospitals
* Intern (DES MBD and ODF).

Exclusion Criteria:

* Students.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: interns + CHU and liberal practitioners; > 160 practitioners
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the state of knowledge relating to the attentional tunnelling of a cohort of odontologists of different professional levels. | At the inclusion
  Face -to-face or online questionnaire (called Attentional Tunnelling in dentistery) including 7 items

SECONDARY OUTCOMES:
Associated risk indicators for attentional tunnelling | At the inclusion
  Face-to-face or online questionnaire (called Attentional Tunnelling) including 2 items. The responses will be given as YES or NO and processed individually (no final score).
Associated risk indicators for prevention strategies | At the inclusion
  Face-to-face or online questionnaire (called Attentional Tunnelling) including 2 items. The responses will be given as YES or NO and processed individually (no final score).
Evaluation of the nature of the means proposed to combat the tunnel effect | At the inclusion
  Online questionnaire including 6 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Dridi, Nice, France